CLINICAL TRIAL: NCT05977543
Title: The Acute Effect of Functional Crackers, Enriched With Grape Seed Flour or With Barley Flour and β-glucans, on Postprandial Glycemic, Lipemic and Antioxidant Metabolism
Brief Title: Acute Effect of Functional Crackers on Postprandial Metabolism
Acronym: Crade23
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of the Aegean (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 12123
Record Dates: First submitted 2023-07-16; First posted 2023-08-04 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: enriched with 10% grape seed flour crackers; 40% barley flour crackers enriched with β-glucan; postprandial effect

STUDY DESIGN:
Intervention Model Description: On enrolment, all subjects were randomly assigned to the C: F1:F2 group (Control: Functional 1: Functional 2), to the F1: C: F2 group (Functional 1: Control: Functional 2) or to the F2: F1: C group (Functional 2: Functional 1: Control). Subjects in the C: F1:F2 group received the Control meal on the first visit, the Functional meal 1 on the second visit and the Functional meal 2 on the third visit; those in the F1:C:F2 group received the Functional meal 1 on the first visit, the Control meal on the second visit and the Functional meal 2 on the third visit while those in the F2:F1:C group received the Functional meal 2 on the first visit, the meal Functional meal 1 on the second visit and the Control meal on the third visit.
Who Masked: Participant
Masking Description: Only investigators knew the group in which each participant were enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control wheat crackers (No Intervention): Volunteers consumed 80g of white bread, 30g of full fat butter and 55g of wheat flour crackers.
- Grape seed flour crackers (Other): Volunteers consumed 80g of white bread, 30g of full fat butter and 55g of wheat flour crackers, enriched with 10% grape seed flour crackers.
  Interventions: Other: Functional crackers enriched with grape seed flour
- Barley flour and β-glucan crackers (Other): Volunteers consumed 80g of white bread, 30g of full fat butter and 55g of 60% wheat flour and 40% barley flour crackers, enriched with β-glucan
  Interventions: Other: Functional crackers with 40% barley flour and enriched with β-glucans

INTERVENTIONS:
Other: Functional crackers enriched with grape seed flour — The crackers was enriched with 10% grape seed flour
  Other Names: Grape seed flour crackers
  Arms: Grape seed flour crackers
Other: Functional crackers with 40% barley flour and enriched with β-glucans — The crackers consisted of 60% wheat flour, 40% barley flour and was enriched with β-glucans.
  Other Names: Barley flour crackers
  Arms: Barley flour and β-glucan crackers

SUMMARY:
The aim of this interventional study was to investigate the postprandial effect of two types of functional crackers, with 10% grape seed flour or 40% barley flour, enriched with β-glucan, in metabolic biomarkers of healthy participants.

DETAILED DESCRIPTION:
A pilot cross-over, controlled, randomized and single-blinded, intervention-clinical trial was carried out, in twelve healthy men and women, aged nineteen to sixty-five years, after random allocation into the control, the grape and the barley interventional groups, received a high-fat and high-carbohydrate meal, containing wheat flour or wheat and 10% grape seed flour or wheat and 40% barley flour, enriched with β-glucan, crackers. Participants consumed the same meals, allocating in cross-over order, with 1 washout week after each trial period. Differences on the metabolism of postprandial serum total, High Density Lipoprotein (HDL-), Low Density Lipoprotein (LDL-) cholesterol, glucose, triglycerides and uric acid levels, as well as of plasma total antioxidant capacity according to Ferric Reducing Antioxidant Power method, were determined between groups in fasting, thirty minutes, one and a half hour, and three hours after meal intake.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-65 years

Exclusion Criteria:

* Age over 65 years old
* History of chronic illness including type I and II diabetes (hemoglobin A1c-HbA1c > 5%)
* Abnormal Body Mass Index (BMI) (>25 kg/m2)
* Alcohol overconsumption (>40 g alcohol/day)
* Abnormal hematological and biochemical profiles (cholesterol > 6.8 mM, triglycerides > 2.8 mM, glucose > 6.11 mM)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Glucose | 3 hours
  Glucose concentration changes from baseline at 3hours
Total Antioxidant Capacity | 3 hours
  Total Antioxidant Capacity concentration changes from baseline at 3 hours

SECONDARY OUTCOMES:
Total cholesterol | 3 hours
  Total cholesterol concentration changes from baseline at 3hours
High Density Lipoprotein cholesterol | 3 hours
  High Density Lipoprotein concentration cholesterol changes from baseline at 3hours
Low Density Lipoprotein cholesterol | 3 hours
  Low Density Lipoprotein cholesterol concentration changes from baseline at 3hours
Triglycerides | 3 hours
  Triglycerides concentration changes from baseline at 3hours
Uric Acid | 3 hours
  Uric Acid concentration changes from baseline at 3hours

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Koutelidakis, Professor, Study Director — University of the Aegean
Locations (1):
- University of the Aegean, Myrina, Limnos/Lesvos, Greece

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data for this study.